CLINICAL TRIAL: NCT02235701
Title: An Open-Label Phase 1/2 Study to Investigate the Preliminary Safety and Activity of Aldoxorubicin Plus Ifosfamide/Mesna in Subjects With Metastatic, Locally Advanced, or Unresectable Soft Tissue Sarcoma
Brief Title: Study to Investigate the Safety and Activity of Aldoxorubicin Plus Ifosfamide/Mesna in Subjects With Metastatic Soft Tissue Sarcoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ImmunityBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALDOXORUBICIN-P1/2-STS-03
Record Dates: First submitted 2014-08-15; First posted 2014-09-10 (Estimated); Results first posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2016-10

CONDITIONS: Metastatic, Locally Advanced, or Unresectable Soft Tissue Sarcoma
Keywords: soft tissue sarcoma; aldoxorubicin; ifosfamide; mesna; phase 1; INNO-206
MeSH Terms: conditions — Neoplasm Metastasis; Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 170 mg/m2 aldoxorubicin (Experimental)
  Interventions: Drug: 170 mg/m2 aldoxorubicin
- 250 mg/m2 aldoxorubicin (Experimental)
  Interventions: Drug: 250 mg/m2 aldoxorubicin

INTERVENTIONS:
Drug: 170 mg/m2 aldoxorubicin — administered at 170 mg/m2 plus 1 gm/m2/day ifosfamide by continuous intravenous infusion for up to 14 days on Day 1 every 28 days
  Arms: 170 mg/m2 aldoxorubicin
Drug: 250 mg/m2 aldoxorubicin — administered at 250 mg/m2 plus 1 gm/m2/day ifosfamide by continuous intravenous infusion for up to 14 days on Day 1 every 28 days
  Arms: 250 mg/m2 aldoxorubicin

SUMMARY:
This is a Phase 1 open-label study to study the safety and activity of aldoxorubicin with ifosfamide/mesna in subjects with metastatic, advanced, unresectable soft tissue sarcoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 15-80 years, male or female.
2. Adjuvant or neoadjuvant chemotherapy (including doxorubicin) allowed if no tumor recurrence for at least 12 months since the last measurement, beginning or end of last chemotherapy.
3. Histologically or cytologically confirmed, locally advanced, unresectable, and/or metastatic soft tissue sarcoma (including rhabdomyosarcoma, Ewing's sarcoma and mixed mesodermal sarcoma), chondrosarcoma or osteosarcoma of intermediate or high grade and gastrointestinal stromal tumors (GIST) (only in subjects that have progressed after receiving treatment with imatinib and sunitinib).
4. Capable of providing informed consent and complying with trial procedures.
5. ECOG performance status 0-2.
6. Life expectancy >12 weeks.
7. Measurable tumor lesions according to RECIST 1.1 criteria.
8. Women must not be able to become pregnant (eg post-menopausal for at least 1 year, surgically sterile, or practicing adequate birth control methods) for the duration of the study. (Adequate contraception includes: oral contraception, implanted contraception, intrauterine device implanted for at least 3 months, or barrier method in conjunction with spermicide.)
9. Males and their female partner(s) of child-bearing potential must use 2 forms of effective contraception (see Inclusion 8 plus condom or vasectomy for males) from the last menstrual period of the female partner during the study treatment and for 6 months after the final dose of study treatment.
10. Women of child bearing potential must have a negative serum or urine pregnancy test at the Screening Visit and be non-lactating.
11. Geographic accessibility to the site that ensures the subject will be able to keep all study-related appointments.

Exclusion Criteria:

1. Prior chemotherapy unless for adjuvant or neoadjuvant therapy with no tumor recurrence for at least 12 months.
2. Prior exposure to >3 cycles or 225 mg/m2 of doxorubicin or Doxil®.
3. Palliative surgery and/or radiation treatment less than 30 days prior to enrollment.
4. Exposure to any investigational agent within 30 days of enrollment.
5. Current Stage 1 or 2 soft tissue sarcomas.
6. Current evidence/diagnosis of alveolar soft part sarcoma, dermatofibrosarcoma, Kaposi's sarcoma, clear cell sarcomas and unresectable low grade liposarcomas.
7. Central nervous system metastasis if symptomatic.
8. History of other malignancies except cured basal cell carcinoma, superficial bladder cancer or carcinoma in situ of the cervix unless documented free of cancer for ≥ 5 years.
9. Laboratory values: Screening serum creatinine >1.5x upper limit of normal (ULN), alanine aminotransferase (ALT) > 3 × ULN or >5 × ULN if liver metastases are present, total bilirubin >3 × ULN, absolute neutrophil count <1,500/mm3, platelet concentration <100,000/mm3, hematocrit level <25% for females or <27% for males, albumin <2 gm/dL, coagulation tests (prothrombin time [PT], partial thromboplastin time [PTT], International Normalized Ratio [INR]) >1.5 × ULN.
10. Clinically evident congestive heart failure > class II of the New York Heart Association (NYHA) guidelines.

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-09-02 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dan Levitt, M.D., Study Director — CytRx Coporation
Locations (1):
- Sarcoma Oncology Center, Santa Monica, California, United States

REFERENCES:
- See also: Related Info — https://doi.org/10.1093/annonc/mdw388.13
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/25312684/

RESULTS

PARTICIPANT FLOW:
Groups:
- 170 mg/m^2 Aldoxorubicin: aldoxorubicin: administered at 170 mg/m^2 plus 1 gm/m2/day ifosfamide by continuous intravenous infusion for up to 14 days on Day 1 every 28 days
- 250 mg/m^2 Aldoxorubicin: aldoxorubicin: administered at 250 mg/m^2 plus 1 gm/m^2/day ifosfamide by continuous intravenous infusion for up to 14 days on Day 1 every 28 days
Period: Overall Study
Arm/Group | 170 mg/m^2 Aldoxorubicin | 250 mg/m^2 Aldoxorubicin
Started | 6 | 64
Completed (Completed defined as receiving at least one dose of study drug.) | 6 | 64
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 170 mg/m^2 Aldoxorubicin: 170 mg/m^2 aldoxorubicin: administered at 170 mg/m^2 plus 1 gm/m^2/day ifosfamide by continuous intravenous infusion for up to 14 days on Day 1 every 28 days
- 250 mg/m^2 Aldoxorubicin: 250 mg/m^2 aldoxorubicin: administered at 250 mg/m^2 plus 1 gm/m^2/day ifosfamide by continuous intravenous infusion for up to 14 days on Day 1 every 28 days
- Total: Total of all reporting groups
Arm/Group | 170 mg/m^2 Aldoxorubicin | 250 mg/m^2 Aldoxorubicin | Total
Number analyzed (Participants) | 6 | 64 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (14.14) | 51.5 (15.05) | 50.5 (15.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 28 | 29
  Male | 5 | 36 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 24 | 25
  Not Hispanic or Latino | 5 | 40 | 45
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 7 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 5 | 56 | 61
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Histologically or cytologically confirmed, locally advanced, unresectable, and/or metastatic STS [Count of Participants; unit: Participants] | 6 | 64 | 70

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events in Participants
Description: The primary objective of this study is to determine the preliminary safety of administration of aldoxorubicin in combination with ifosfamide in subjects with metastatic, locally advanced, or unresectable soft tissue sarcoma as measured by the frequency and severity of adverse events (AEs).
  The following assessments were used to determine if subjects had adverse events:
  * vitals signs (systolic/diastolic blood pressure, pulse, respiration, temperature, weight, and body surface area)
  * physical examination
  * laboratory tests (chemistry, hematology, urinalysis, anion gap)
  additionally, the following scans were performed to determine adverse events:
  * ECHO / MUGA
  * ECG
Time Frame: Treatment was planned to continue until tumor progression is observed, subject asks to withdraw, or unacceptable toxicity occurs (up to 766 days).
Measure: Count of Participants; unit: Participants
Groups:
- 170 mg/m^2 Aldoxorubicin: aldoxorubicin: administered at 170 mg/m^2 plus 1 gm/m^2/day ifosfamide by continuous intravenous infusion for up to 14 days on Day 1 every 28 days
Arm/Group | 170 mg/m^2 Aldoxorubicin | 250 mg/m^2 Aldoxorubicin
Number analyzed (Participants) | 6 | 64
Participants | 6 | 64

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) that occurred after any administration of the study medication were to be followed until the event resolved, or until 30 days after the last dose of study medication. All SAEs that occurred during the course of the study or within 30 days of the last administration of study medication were to be reported, up to 766 days.
Groups:
- 250 mg/m^2 Aldoxorubicin: aldoxorubicin: administered at 250 mg/m^2 plus 1 gm/m2/day ifosfamide by continuous intravenous infusion for up to 14 days on Day 1 every 28 days
Arm/Group | 170 mg/m^2 Aldoxorubicin | 250 mg/m^2 Aldoxorubicin
All-Cause Mortality (participants affected / at risk) | 0/6 | 16/64
Serious Adverse Events (participants affected / at risk) | 3/6 | 31/64
Other Adverse Events (participants affected / at risk) | 6/6 | 64/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 170 mg/m^2 Aldoxorubicin (N=6) | 250 mg/m^2 Aldoxorubicin (N=64)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 8
Anemia (Blood and lymphatic system disorders) | 0 | 6
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Ophthalmoplegia (Eye disorders) | 0 | 1
Small bowel obstruction (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
Pyrexia (General disorders) | 0 | 3
Asthenia (General disorders) | 0 | 1
Systemic inflammatory response syndrome (General disorders) | 0 | 1
Enterobacter Bacteremia (Infections and infestations) | 1 | 0
Enterobacter sepsis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 4
Urinary tract infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Klebsiella bacteremia (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 2
Device related sepsis (Infections and infestations) | 0 | 1
Viral syndrome (Infections and infestations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Tumor necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Sarcomatosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 0 | 1
Neurotoxicity (Nervous system disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypertension (Vascular disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Cellulitis of male external genitalia (Infections and infestations) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Wound necrosis (Injury, poisoning and procedural complications) | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 170 mg/m^2 Aldoxorubicin (N=6) | 250 mg/m^2 Aldoxorubicin (N=64)
Anaemia (Blood and lymphatic system disorders) | 6 | 56
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 9
Leukopenia (Blood and lymphatic system disorders) | 1 | 6
Neutropenia (Blood and lymphatic system disorders) | 6 | 60
Splenomegaly (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 29
Tachycardia (Cardiac disorders) | 1 | 8
Abdominal pain (Gastrointestinal disorders) | 0 | 7
Constipation (Gastrointestinal disorders) | 2 | 11
Dyspepsia (Gastrointestinal disorders) | 0 | 4
Nausea (Gastrointestinal disorders) | 4 | 45
Stomatitis (Gastrointestinal disorders) | 0 | 10
Vomiting (Gastrointestinal disorders) | 1 | 28
Fatigue (General disorders) | 6 | 52
Oedema Peripheral (General disorders) | 0 | 5
Pyrexia (General disorders) | 1 | 13
Hypoalbuminaemia (Hepatobiliary disorders) | 1 | 0
Enterobacter Bacteraemia (Infections and infestations) | 1 | 0
Enterobacter Sepsis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 5
Upper respiratory tract infection (Infections and infestations) | 1 | 3
Staphylococcal infection (Infections and infestations) | 2 | 2
Varicella zoster virus infection (Infections and infestations) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 7
Alanine aminotransferase increased (Investigations) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 7
Dehydration (Metabolism and nutrition disorders) | 0 | 8
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 8
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 20
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 7
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 3
Neurotoxicity (Nervous system disorders) | 0 | 4
Anxiety (Psychiatric disorders) | 0 | 10
Insomnia (Psychiatric disorders) | 0 | 12
Dysuria (Renal and urinary disorders) | 0 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 12
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 5
Deep vein thrombosis (Vascular disorders) | 0 | 4
Hypotension (Vascular disorders) | 1 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-30): https://cdn.clinicaltrials.gov/large-docs/01/NCT02235701/Prot_SAP_000.pdf